CLINICAL TRIAL: NCT06243484
Title: Clinical Study to Investigate the Effect of the Food Supplement TOTUM-070 on Lipid Metabolism in Moderately Hypercholesterolemic Subjects After 3 Months of Supplementation
Brief Title: Effect of the Food Supplement TOTUM-070 on Lipid Metabolism
Acronym: HEARTII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VCT-013; BTS1876_22 (Other: Biotesys)
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: A MULTICENTER, RANDOMIZED PLACEBO-CONTROLLED DOUBLE-BLINDED STUDY
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted in a double-blind randomized manner. The random allocation sequence will be provided sealed to the independent pharmacist (not involved in the study) by an independent statistician. The ratio of randomization between the verum and placebo groups will be 1:1. Stratification randomization will be performed according to LDL-c at V0 (<160 mg/dL / ≥ 160 mg/dL) and site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOTUM-070 (Experimental): The experimental arm will be supplemented with TOTUM-070 twice a day
  Interventions: Dietary Supplement: TOTUM-070
- PLACEBO (Placebo Comparator): The placebo comparator arm will be supplemented with a placebo twice a day
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: TOTUM-070 — 12 weeks of TOTUM-070 supplementation with Placebo (blinded arms)
  Other Names: Active product 2 intakes per day
  Arms: TOTUM-070
Dietary Supplement: PLACEBO — 8 capsules per day to consume orally in two intakes
  Other Names: Comparator product 2 intakes per day
  Arms: PLACEBO

SUMMARY:
This clinical trial is to confirm the effects of TOTUM-070, a mix of 5 plants extracts, consumed at the daily regimen of two times per day, on fasting blood LDL cholesterol concentrations in moderately hypercholesterolemic subjects after 12 weeks of consumption (V3).

DETAILED DESCRIPTION:
The main objective is to confirm the efficacy of a 4.995g/day dose of TOTUM-070 versus placebo on fasting blood LDL cholesterol level (Ultracentrifugation (UC) method) in moderately hypercholesterolemic subjects following 12 weeks of consumption (V3).

The proposed double-blinded, placebo-controlled, clinical study will provide further insight into the safety and efficacy of TOTUM-070 at the same dose (4.995g/day) on a shorter supplementation period (3 months) than the previous one (6 months), as well as assess the effect after the follow-up period without product intake.

ELIGIBILITY:
Main Inclusion Criteria:

* I1. From 18 to 70 years (including ranges);
* I2. BMI of ≥18.5 and ≤35 kg/m²;
* I3. Moderately hypercholesterolemic subject without any clinical symptoms of hypercholesterolemia (xanthoma, recurrent chest and/or leg pain…) and not requiring immediate pharmacological lipid-lowering treatment;
* I4. Weight stable within ± 5% in the last three months before V0;
* I5. SCORE2 - SCORE2-OP (Older Persons) Cardiovascular Risk Chart

Main Exclusion Criteria:

* E1. Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal dysfunction or other metabolic disorder needing a dose adjustment in drug intervention according to the professional recommendations;
* E2. Suffering from an uncontrolled arterial hypertension;
* E3. With a history of ischemic cardiovascular event;
* E4. Having undergone recent surgical procedure in the past 6 months before V0 or planned in the 5 months to come;
* E5. History of bariatric surgery;
* E6. Suffering from a severe chronic disease;
* E7. For women: ongoing pregnancy (as evidenced by a positive test for β-Human Chorionic Gonadotropin, i.e. > 5 mUI/mL, realized at V0) or breastfeeding or finished since less than 6 months before V0 or intending to become pregnant within 5 months ahead;
* E8. Under cholesterol and/or lipid-lowering treatment or stopped less than 3 months before the inclusion visit V0;
* E9. Under medication which could affect blood lipid parameters or stopped less than 3 months before the inclusion visit V0 (antihypertensive stable long-term treatment tolerated);
* E10. Consuming more than 3 standard drinks daily of alcoholic beverage for men or 2 standard drinks daily for women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of fasting blood LDL cholesterol level | Baseline (V1) and End of consumption after 12 weeks (V3)
  Fasting blood LDL cholesterol level by Ultracentrifugation method

SECONDARY OUTCOMES:
Evolution of fasting blood LDL cholesterol level | Baseline (V1), Following 6 weeks of consumption (V2) and 6 weeks after the end of consumption (V4)
  Fasting blood LDL cholesterol level by Ultracentrifugation method
Evolution of Lipid profile | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Triglycerides, Total-cholesterol, HDL-C, non-HDL-C, LDL-C, Free Fatty Acids, Apo-A1 and Apo-B, Apo-B/Apo-A1 ratio, Apo-C3
Evolution of Lipid homeostasis indices | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Atherogenic index (ratio of triglycérides and HDL-C), atherogenic coefficient (ratio of total-cholesterol and HDL-C), cardiac risk ratio 1 (ratio of total-cholesterol and HDL-C), cardiac risk ratio 2 (ratio of LDL-C and HDL-C) (note that all these measures are unitless ratios)
Evolution of fasting glycemia | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Fasting Glycemia (in mg/dL)
Evolution of Low grade inflammation | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Fasting blood hsCRP, Interleukin-6
Evolution of body weight | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Body weight (BW) in kg
Evolution of body mass index | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Body mass index (BMI) in kg/m2
Evolution of waist circumference | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Waist circumference (WC) in cm
Evolution of hip circumference | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Hip circumference (HC) in cm
Evolution of waist to hip ratio | Baseline (V1), Following 6 weeks of consumption (V2), at the end of consumption after 12 weeks (V3) and 6 weeks after the end of consumption (V4)
  Waist to hip ratio (WHR)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — Biotesys
Locations (1):
- Biotesys, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No